CLINICAL TRIAL: NCT02513537
Title: Postoperative Delirium - European Society of Anaesthesiology Survey
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: PODESAS
Record Dates: First submitted 2015-03-20; First posted 2015-07-31 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The ESA is currently preparing a guideline on the management of postoperative delirium (POD), which attempts to reduce the impact of postoperative delirium and provide recommendations for prevention, diagnostics and treatment of delirium outside the intensive care unit. The guidelines are going to be published during 2015.

While the guideline provides recommendations for daily practice, assessment of current practice and knowledge is of utmost importance, because the implementation and the measurement of a change in clinical practice will be dependent on these measurements.

This Survey has been approved by the Scientific and Research Committees of the European Society of Anaesthesiology (ESA), the Media Committee of the ESA, as well as the institutional ethical committee of Charité - Universitätsmedizin Berlin.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesists, nursing staff, which are invited to the online - Survey of the European Society of Anaesthesiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anaesthesists , nursing statt and students (Members of the European Society of Anaesthesiology)
Sampling Method: Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2015-08; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Status of diagnosis of delirium | Up to 6 months
  Answers of ESA-members regarding diagnosis instruments of Delirium. Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non mandatory).
Status of prevention of delirium | Up to 6 months
  Answers of ESA-members regarding prevention measurements of Delirium Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non mandatory).
Status of therapy of delirium | Up to 6 months
  Answers of ESA-members regarding therapy of Delirium. Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non-mandatory).

SECONDARY OUTCOMES:
Status of diagnosis of delirium | Up to one, two and five years
  Answers of ESA-members regarding diagnosis instruments of Delirium. Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non-mandatory).
Status of prevention of delirium | Up to one, two and five years
  Answers of ESA-members regarding prevention measurements of Delirium. Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non-mandatory).
Status of therapy of delirium | Up to one, two and five years
  Answers of ESA-members regarding therapy of Delirium. Survey: Multiple Chioce Question. Plus short Essay question to describe prevention (non-structured, non-mandatory).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité - Univeristy Medicine Berlin
Locations (4):
- Department of Anaesthesiolgy and Intensive Care Medicine CVK/CCM, Charité - Univeristy Medicine Berlin, Berlin, Germany
- Italian National Research Centres On Aging, Ancona, Italy
- Department of Anaesthesiology, Faculdad de medicina de Valladloid, Hospital Universitario Rio Hortega, Valladolid, Spain
- Department of Anaesthesia, Imperial College NHS Healthcare Trust, London, United Kingdom